CLINICAL TRIAL: NCT06808607
Title: Thrombotic Outcome of Primary Versus Secondary Antiphospholipid Syndrome
Brief Title: Clinical Outcomes of Primary Versus Secondary Antiphospholipid Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Mohammed Abdel-Aziz, Lecturer of Clinical Hematology, Faculty of medicine, Assiut university, Assiut University
Other Study IDs: 04-2024-300543
Record Dates: First submitted 2025-01-12; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Antiphospholipid Syndrome
Keywords: Thrombosis; Antiphospholipid syndrome
MeSH Terms: conditions — Antiphospholipid Syndrome; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective to compare clinical outcomes of primary versus secondary antiphospholipi: Observational study to compare clinical outcomes of primary versus secondary antiphospholipid syndrome

SUMMARY:
Observational retrospective cohort study to assess clinical outcomes in patients with primary versus secondary antiphospholipid syndrome

DETAILED DESCRIPTION:
Antiphospholipid antibody syndrome is an autoimmune disorder associated with positive antiphospholipid antibodies including the lupus anticoagulant, anticardiolipin antibodies IgG or IgM, and/or anti-ß2-glycoprotein IgG or IgM associated with thrombotic problems and pregnancy loss.

Antiphospholipid syndrome is one of the most frequent forms of acquired thrombophilia and is associated with an increased risk of both venous and arterial thrombotic events. Thirty to 40% of systemic lupus erythematosus (SLE) patients have associated antiphospholipid syndrome.

Antiphospholipid syndrome has estimated incidence in the general population of 2.1 (1.4-2.8) per 100 000, and the prevalence of 50 (42-58) per 100 000. APS is more common in female with a female to male ratio is 3.5:1 for primary and 7:1 for secondary.

Antiphospholipid syndrome is divided into two types primary syndrome without an underlying disease, and secondary antiphospholipid syndrome that is associated with another autoimmune syndrome, most commonly Systemic Lupus Erythematosus (SLE).

Patients with APS are more at risk of recurrent thrombosis (3). n a retrospective analysis of 160 patients with APS, venous thromboembolism (VTE) was found to be the commonest manifestation (47.5%) followed by arterial thromboembolism (43.1%) then materno fetal problems which were found only in 9.7% of patients, and finally, catastrophic antiphospholipid syndrome (CAPS) represented in only 2.5 percent of the cases (4).

The clinical manifestations of antiphospholipid syndrome include haematological (thrombocytopenia, venous thrombosis), obstetrical (recurrent pregnancy loss), neurological (stroke, transient ischaemic attack, seizures), cardiovascular, dermatological such as livedo reticularis, skin ulceration and necrosis, renal (glomerulonephritis and renal thrombotic microangiopathy), and orthopedic (avascular necrosis of bones).

the manifestation spectrum ranged from asymptomatic antiphospholipid antibodies positivity, various non-criteria manifestations, obstetric morbidity, thrombosis, to life-threatening catastrophic antiphospholipid syndrome. The wide manifestation spectrum led to a heterogeneous entity and brought challenges to management of the syndrome.

The aim of this study was to compare primary versus secondary effects of antiphospholipid syndrome on the development of thrombosis and its outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed as antiphospholipid syndrome in clinical hematology or rheumatology units in internal medicine department, Assiut university hospital.

Exclusion Criteria:

* patients with other risk factor for thrombosis (malignancy, cocs, protein c or protein s deficiency etc

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Retrospective cohort
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-02-07 (Estimated); Primary Completion 2026-03-06 (Estimated); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
to compare percentage of patients with primary versus secondary antiphospholipid syndrome in developing recurrent thrombosis | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Maha Abdel-Aziz, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Undecided yet

REFERENCES:
- See also: Related Info — https://doi.org/10.1186/s13075-022-02814-w
- See also: Related Info — https://doi.org/10.1016/j.ejr.2022.11.002
- See also: Related Info — https://doi.org/10.1016/j.jaut.2018.05.007